CLINICAL TRIAL: NCT01582958
Title: The Effect of Osteopathic Manipulative Treatment on Patients With Chronic Obstructive Pulmonary Disease:Correlating Pulmonary Function Tests With Biochemical Alterations
Brief Title: The Effect of OMT on Patients With COPD: Correlating Pulmonary Function Tests With Biochemical Alterations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Sherman Gorbis, DO, FAAO, Principal Investigator, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122470
Record Dates: First submitted 2012-04-14; First posted 2012-04-23 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Osteopathic Manipulative Treatment; Pulmonary Function Tests; Biochemical Alterations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment (Experimental): This arm will receive the usual Pulmonary Rehabilitation Program plus OMT, the intervention.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)
- placebo (Placebo Comparator): Receives normal pulmonary rehabilitation care plus positioned to receive OMT but OMT is not provided.
  Interventions: Other: sham omt
- Control (No Intervention): This arm receives only pulmonary rehabilitation care.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — Osteopathic Manipulative Treatment (OMT) is the therapeutic application of manually guided forces by an Osteopathic physician to improve physiologic function.
  Other Names: Other names are not applicable.
  Arms: Treatment
Other: sham omt — Hands are placed on subjects the same as omt arm but no omt is provided.
  Other Names: Other names are not applicable.
  Arms: placebo

SUMMARY:
This project proposes to test the hypothesis that osteopathic manipulative treatment (OMT) given to patients with moderate to severe chronic obstructive pulmonary disease (COPD) enrolled in a 12-week pulmonary rehabilitation program (PRP) will result in improved respiratory pump function over and above that seen in sham and control groups. Specifically, we will study the effects of three OMT techniques: (a) thoracic inlet indirect myofascial release; (b) rib raising with continued stretch of the paraspinal muscle to the L2 level; and (c) cervical paraspinal muscle stretch with suboccipital muscle release. The key clinical readouts will include: spirometry, P100 (and index of diaphragm and inspiratory muscle efficiency), maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP), as well as laser evaluation of chest wall excursion. Supplementing these objective parameters will be several more subjective clinical outcome measures: exercise tolerance (6-minute walk test), dyspnea (shortness of breath questionnaire), and quality of life questionnaire. Finally, an attempt will be made to correlate biochemical alterations that may shed light on the biological mechanism underlying the OMT procedures.

DETAILED DESCRIPTION:
According to the above directions (provide a more extensice description, if desired), I am choosing to just submit the brief summary.

Thank you, Sherman Gorbis, DO

ELIGIBILITY:
Inclusion Criteria:

* postbronchodilator FEV1/FVC <0.7 and FEV1 <80% predicted [FEV1 =volume that has been exhaled at the end of the first second of forced expiration] and FVC volume of air that can be forcibly blown out after full inspiration]
* history of smoking >20 pack-years
* stable condition at inclusion with no infection or exacerbation for at least two months
* optimal medical therapy for at least eight weeks with no change

Exclusion Criteria:

* history of active pulmonary disease such as asthma
* positive bronchodilator test
* treatment with N-acetylcysteine
* previous diagnosis of hypertension or current anti-hypertensive treatment
* known unstable or moderate to severe heart disease (arrhythmia, ischemic heart disease, or cardiomyopathy)
* previous diagnosis of chronic illness such as diabetes, renal failure, hypercholesterolemia, hepatic cirrhosis, cancer, rheumatoid arthritis or any other systemic inflammatory disease
* neuromuscular or disabling cognitive problems
* engagement in any exercise-training program during the past three months
* substance abuse in the preceding six months

Ages: 49 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in spirometry at 6 weeks and 12 weeks | baseline, 6 weeks, 12 weeks
  amount (volume) and/or speed (flow) of air that can be inhaled and exhaled
Change from baseline in P100 at 6 weeks and 12 weeks | baseline, 6 weeks, 12 weeks
  an index of diaphragm and inspiratory muscle efficiency (endurance)
Change from baseline in MIP (maximum inspiratory pressure) and MEP (maximum expiratory pressure)at 6 weeks and 12 weeks. | baseline, 6 weeks, 12 weeks
  assessments of inspiratory and expiratory muscle function, respectively
Change from baseline in inspiratory capacity at 6 weeks and 12 weeks. | baseline, 6 weeks, 12 weeks
  representing an indirect evaluation of chest wall excursion

SECONDARY OUTCOMES:
Change from baseline in exercise tolerance at 6 weeks and 12 weeks. | baseline, 6 weeks, 12 weeks
  6-minute walk test
Change from baseline in dyspnea (shortness of breath) at 6 weeks and 12 weeks. | baseline, 6 weeks, 12 weeks
  shortness of breath questionnaire
Change from baseline in quality of life at 6 weeks and 12 weeks. | baseline, 6 weeks, 12 weeks
  Short Form 36 questionnaire
Change from baseline in profiling of the plasma metabolome at 6 weeks and 12 weeks. | baseline, 6 weeks, 12 weeks
  mass spectrometry (both non-targeted profiling of entire suite of metabolites and targeted profiling of oxylipins and endocannabinoid metabolites
Change from baseline in profiling of plasma proteins at 6weeks and 12 weeks. | baseline, 6 weeks, 12 weeks
  antibody microarray analysis (particularly targeting the inflammatory/anti-inflammatory cytokines)

CONTACTS AND LOCATIONS:
Overall Officials: Sherman Gorbis, DO, Principal Investigator — Michigan State University
Locations (1):
- McClaren Greater Lansing, Lansing, Michigan, United States